CLINICAL TRIAL: NCT03767374
Title: Risk-factors for Multidrug-resistant (MDR) and Extensively Drug-resistant (XDR) Bacteria Colonization Among Patients at High Risk of STIs
Brief Title: Risk-factors for Multidrug-resistant Bacteria Colonization Among Patients at High Risk of STIs
Acronym: BMR-IST
Status: Completed | Type: Observational
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: IMEA 52
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2022-10

CONDITIONS: Bacterial Infections; HIV Infections
Keywords: MDR, XDR, ESBL, ESBL, MRSA, CRE; HIV, PrEP, CeGIDD, STI, bacteria colonization
MeSH Terms: conditions — Bacterial Infections; HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Inguinal (at inclusion) and anal swab samples (at inclusion and after 6 months) Fecal sample (at inclusion and after 6 months, only for patients identified with ESBL and/or CRE colonization)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main study group (HIV-negative): 2000 HIV-negative individuals seeking care at the STI clinic of Saint-Antoine Hospital
  * Inguinal swab sample
  * Anal swab sample
  * Fecal sample
  * Risk factor assessment
  Interventions: Procedure: Inguinal swab sample; Procedure: Anal swab sample; Procedure: Fecal sample; Other: Risk factor assessment
- Exposure-matched group (HIV-positive): 500 HIV-positive men who have sex with men from the Infectious Diseases Unit of Saint- Antoine Hospital. These individuals will be compared to 500 HIV-negative MSM from the main study group, matching on age (+/-5 years).
  * Inguinal swab sample
  * Anal swab sample
  * Fecal sample
  * Risk factor assessment
  Interventions: Procedure: Inguinal swab sample; Procedure: Anal swab sample; Procedure: Fecal sample; Other: Risk factor assessment

INTERVENTIONS:
Procedure: Inguinal swab sample — Inguinal samples using swab at cross-sectional visit
  Other Names: ESwab
Procedure: Anal swab sample — Anal samples using swab at cross-sectional visit and at 6-month visit (for those with ESBL and/or CRE colonization)
  Other Names: ESwab
Procedure: Fecal sample — Fecal sample at cross-sectional visit and at 6-month visit (for those with ESBL and/or CRE colonization)
Other: Risk factor assessment — Patients will be asked questions on risk factors associated with MDR/XDR colonization at cross-sectional visit and at 6-month visit (for those with ESBL and/or CRE colonization

SUMMARY:
The aim of this study is to identify risk factors and prevalence of multidrug-resistant (MDR) and extensively drug-resistant (XDR) bacteria colonization among patients at high risk of STIs

DETAILED DESCRIPTION:
The spread of multidrug-resistant (MDR) and extensively drug-resistant (XDR) bacteria have become a worldwide public health concern. Infection with MDR/XDR bacteria is associated with increased morbidity, increased risk of therapeutic failure and healthcare costs. The largest burden is from extended-spectrum betalactamase-producing enterobacteriaceae (ESBL) and carbapenem-resistant enterobacteriaceae (CRE).

The World Health Organization (WHO) has considered the epidemic of MDR/XDR bacteria as a major health concern and has registered these bacteria in the "priory pathogens list." This list includes pathogens for which new antibiotics are urgently needed. Moreover, in their recent report on ESBL, the French National Authorities of Health (HAS) has recommended that additional studies be conducted to improve knowledge about colonization risk factors.

Some risk factors have been already identified: antibiotic intake and travel to countries with high MCR/XDR bacteria prevalence; however, many others are poorly identified. Patients visiting the CeGIDD (free information, screening and diagnosis center for sexually transmitted infections) and those receiving pre-exposure prophylaxis (PrEP) to prevent HIV infection are more exposed to STIs (including methicillin-resistant staphylococcus aureus, MRSA) and receive antibiotics for STI treatment. Moreover, an increase of STIs has been recently observed in men who have sex with men and in patients receiving PrEP. As antibiotic use is likely considerably increased in this population, we anticipate a high proportion with MDR/XDR colonization.

The objective of the "BMR-IST" study is to identify risk-factors (i.e. sexual behaviors, HIV status, antiretroviral PrEP, STIs, antibiotic use and travel to epidemic countries) of MDR/XDR bacteria colonization among patients at high risk of acquiring STIs and to determine the prevalence of MDR colonization in the studied population.

ELIGIBILITY:
Cohort 1 -

Inclusion Criteria:

* Age ≥ 18 years
* Consulting at the STI clinic of Saint-Antoine Hospital
* Signed the informed consent form

Non-inclusion criteria:

- No fluency in French

Cohort 2 -

Inclusion criteria:

* Men who have sex with men
* Seeking care at Saint-Antoine Hospital
* HIV-positive

Non-inclusion criteria:

- No fluency in French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1: HIV-negative individuals at high risk of STI infection seeking care at a STI testing center in Paris, France
  Cohort 2: HIV-positive individuals seeking care at a university hospital in Paris, France
Sampling Method: Non-Probability Sample
Enrollment: 2186 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of ESBL and/or CRE colonization | 0 months
  Proportion of participants with ESBL and/or CRE colonization

SECONDARY OUTCOMES:
Loss of ESBL and/or CRE colonization after 6 months | 6 months
  Proportion of ESBL and/or CRE colonized participants no longer colonized at 6 months
STI prevalence | 0 months
  Proportion of participants with an STIs
Prevalence of ESBL and/or CRE colonization in the HIV-negative MSM group | 0 months
  Proportion of HIV-negative MSM participants with ESBL and/or CRE colonization
Prevalence of ESBL and/or CRE colonization in the HIV-positive MSM group | 0 months
  Proportion of HIV-positive MSM participants with ESBL and/or CRE colonization
Prevalence of ESBL and/or CRE colonization in the PrEP group | 0 months
  Proportion of participants undergoing PrEP with ESBL and/or CRE colonization
Prevalence of ESBL and/or CRE colonization in those with previous antibiotic exposure | 0 months
  Proportion of participants having previous antibiotic exposure with ESBL and /or CRE colonization

CONTACTS AND LOCATIONS:
Overall Officials: Laure Surgers, MD, Principal Investigator — Saint-Antoine Hospital, Paris, France 75012
Locations (1):
- CeGIDD and Infections Diseases Unit, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided later by the scientific committee at the end of the study.

REFERENCES:
- [Background] Ben-Ami R, Rodriguez-Bano J, Arslan H, Pitout JD, Quentin C, Calbo ES, Azap OK, Arpin C, Pascual A, Livermore DM, Garau J, Carmeli Y. A multinational survey of risk factors for infection with extended-spectrum beta-lactamase-producing enterobacteriaceae in nonhospitalized patients. Clin Infect Dis. 2009 Sep 1;49(5):682-90. doi: 10.1086/604713. PMID 19622043
- [Background] Canton R, Coque TM. The CTX-M beta-lactamase pandemic. Curr Opin Microbiol. 2006 Oct;9(5):466-75. doi: 10.1016/j.mib.2006.08.011. Epub 2006 Aug 30. PMID 16942899
- [Background] Coque TM, Baquero F, Canton R. Increasing prevalence of ESBL-producing Enterobacteriaceae in Europe. Euro Surveill. 2008 Nov 20;13(47):19044. PMID 19021958
- [Background] Diep BA, Chambers HF, Graber CJ, Szumowski JD, Miller LG, Han LL, Chen JH, Lin F, Lin J, Phan TH, Carleton HA, McDougal LK, Tenover FC, Cohen DE, Mayer KH, Sensabaugh GF, Perdreau-Remington F. Emergence of multidrug-resistant, community-associated, methicillin-resistant Staphylococcus aureus clone USA300 in men who have sex with men. Ann Intern Med. 2008 Feb 19;148(4):249-57. doi: 10.7326/0003-4819-148-4-200802190-00204. Epub 2008 Jan 30. PMID 18283202
- [Background] Gaudreau C, Pilon PA, Sylvestre JL, Boucher F, Bekal S. Multidrug-Resistant Campylobacter coli in Men Who Have Sex with Men, Quebec, Canada, 2015. Emerg Infect Dis. 2016 Sep;22(9):1661-3. doi: 10.3201/eid2209.151695. No abstract available. PMID 27533504
- [Background] Harris AD, McGregor JC, Johnson JA, Strauss SM, Moore AC, Standiford HC, Hebden JN, Morris JG Jr. Risk factors for colonization with extended-spectrum beta-lactamase-producing bacteria and intensive care unit admission. Emerg Infect Dis. 2007 Aug;13(8):1144-9. doi: 10.3201/eid1308.070071. PMID 17953083
- [Background] Jean SS, Lee WS, Lam C, Hsu CW, Chen RJ, Hsueh PR. Carbapenemase-producing Gram-negative bacteria: current epidemics, antimicrobial susceptibility and treatment options. Future Microbiol. 2015;10(3):407-25. doi: 10.2217/fmb.14.135. PMID 25812463
- [Background] Livermore DM, Canton R, Gniadkowski M, Nordmann P, Rossolini GM, Arlet G, Ayala J, Coque TM, Kern-Zdanowicz I, Luzzaro F, Poirel L, Woodford N. CTX-M: changing the face of ESBLs in Europe. J Antimicrob Chemother. 2007 Feb;59(2):165-74. doi: 10.1093/jac/dkl483. Epub 2006 Dec 6. PMID 17158117
- [Background] Livermore DM. Has the era of untreatable infections arrived? J Antimicrob Chemother. 2009 Sep;64 Suppl 1:i29-36. doi: 10.1093/jac/dkp255. PMID 19675016
- [Background] Molina JM, Capitant C, Spire B, Pialoux G, Cotte L, Charreau I, Tremblay C, Le Gall JM, Cua E, Pasquet A, Raffi F, Pintado C, Chidiac C, Chas J, Charbonneau P, Delaugerre C, Suzan-Monti M, Loze B, Fonsart J, Peytavin G, Cheret A, Timsit J, Girard G, Lorente N, Preau M, Rooney JF, Wainberg MA, Thompson D, Rozenbaum W, Dore V, Marchand L, Simon MC, Etien N, Aboulker JP, Meyer L, Delfraissy JF; ANRS IPERGAY Study Group. On-Demand Preexposure Prophylaxis in Men at High Risk for HIV-1 Infection. N Engl J Med. 2015 Dec 3;373(23):2237-46. doi: 10.1056/NEJMoa1506273. Epub 2015 Dec 1. PMID 26624850
- [Background] Landry MM, Sarma DP. In-situ chondrosarcoma of the foot arising in a solitary enchondroma. J Foot Surg. 1990 Jul-Aug;29(4):324-6. PMID 2229904
- [Background] Nicolas-Chanoine MH, Gruson C, Bialek-Davenet S, Bertrand X, Thomas-Jean F, Bert F, Moyat M, Meiller E, Marcon E, Danchin N, Noussair L, Moreau R, Leflon-Guibout V. 10-Fold increase (2006-11) in the rate of healthy subjects with extended-spectrum beta-lactamase-producing Escherichia coli faecal carriage in a Parisian check-up centre. J Antimicrob Chemother. 2013 Mar;68(3):562-8. doi: 10.1093/jac/dks429. Epub 2012 Nov 9. PMID 23143897
- [Background] Osthoff M, McGuinness SL, Wagen AZ, Eisen DP. Urinary tract infections due to extended-spectrum beta-lactamase-producing Gram-negative bacteria: identification of risk factors and outcome predictors in an Australian tertiary referral hospital. Int J Infect Dis. 2015 May;34:79-83. doi: 10.1016/j.ijid.2015.03.006. Epub 2015 Mar 11. PMID 25769526
- [Background] Rodriguez-Bano J, Lopez-Cerero L, Navarro MD, Diaz de Alba P, Pascual A. Faecal carriage of extended-spectrum beta-lactamase-producing Escherichia coli: prevalence, risk factors and molecular epidemiology. J Antimicrob Chemother. 2008 Nov;62(5):1142-9. doi: 10.1093/jac/dkn293. Epub 2008 Jul 18. PMID 18641033
- [Background] Ruppe E, Lixandru B, Cojocaru R, Buke C, Paramythiotou E, Angebault C, Visseaux C, Djuikoue I, Erdem E, Burduniuc O, El Mniai A, Marcel C, Perrier M, Kesteman T, Clermont O, Denamur E, Armand-Lefevre L, Andremont A. Relative fecal abundance of extended-spectrum-beta-lactamase-producing Escherichia coli strains and their occurrence in urinary tract infections in women. Antimicrob Agents Chemother. 2013 Sep;57(9):4512-7. doi: 10.1128/AAC.00238-13. Epub 2013 Jul 8. PMID 23836184
- [Background] Schwaber MJ, Navon-Venezia S, Kaye KS, Ben-Ami R, Schwartz D, Carmeli Y. Clinical and economic impact of bacteremia with extended- spectrum-beta-lactamase-producing Enterobacteriaceae. Antimicrob Agents Chemother. 2006 Apr;50(4):1257-62. doi: 10.1128/AAC.50.4.1257-1262.2006. PMID 16569837
- [Background] Szumowski JD, Wener KM, Gold HS, Wong M, Venkataraman L, Runde CA, Cohen DE, Mayer KH, Wright SB. Methicillin-resistant Staphylococcus aureus colonization, behavioral risk factors, and skin and soft-tissue infection at an ambulatory clinic serving a large population of HIV-infected men who have sex with men. Clin Infect Dis. 2009 Jul 1;49(1):118-21. doi: 10.1086/599608. PMID 19480576
- [Background] Tumbarello M, Sanguinetti M, Montuori E, Trecarichi EM, Posteraro B, Fiori B, Citton R, D'Inzeo T, Fadda G, Cauda R, Spanu T. Predictors of mortality in patients with bloodstream infections caused by extended-spectrum-beta-lactamase-producing Enterobacteriaceae: importance of inadequate initial antimicrobial treatment. Antimicrob Agents Chemother. 2007 Jun;51(6):1987-94. doi: 10.1128/AAC.01509-06. Epub 2007 Mar 26. PMID 17387156
- [Background] Woerther PL, Burdet C, Chachaty E, Andremont A. Trends in human fecal carriage of extended-spectrum beta-lactamases in the community: toward the globalization of CTX-M. Clin Microbiol Rev. 2013 Oct;26(4):744-58. doi: 10.1128/CMR.00023-13. PMID 24092853